CLINICAL TRIAL: NCT07043972
Title: Phase II Study of Second-line Gemcitabine Plus Carboplatin After Progression on Enfortumab Vedotin With Pembrolizumab in Advanced or Metastatic Urothelial Carcinoma
Brief Title: Gemcitabine and Carboplatin After Progression on Enfortumab Vedotin and Pembrolizumab in Advanced/Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-230; 25-1008 (Other: IRB)
Record Dates: First submitted 2025-06-26; First posted 2025-06-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma
Keywords: phase II; locally advanced urothelial cancer; gemcitabine plus carboplatin; enfortumab vedotin plus pembrolizumab; metastatic urothelial cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine plus carboplatin (Experimental): Patients will be treated with gemcitabine 1,000 mg/m2 administered over 30 minutes IV on days 1 and 8, followed by carboplatin area under the curve (AUC) 5 on day 1, every 3 weeks.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Gemcitabine — IV over 30 minutes given on days 1 and 8 of a 21 day cycle
Drug: Carboplatin — IV over 30 minutes given on day 1 of a 21 day cycle

SUMMARY:
The goal of this clinical trial is to learn if a chemotherapy combination called gemcitabine and carboplatin (GC) works to treat advanced urothelial cancer in people who have already been treated with enfortumab vedotin and pembrolizumab (EVP).

It will also learn about the efficacy and safety of GC in these patients.

The main questions it aims to answer are:

* Does GC shrink the cancer or stop it from growing?
* What medical side effects do participants have while receiving GC?

Researchers will study how GC affects survival, cancer control, and quality of life. They will also collect blood samples to look at health-related markers and cancer DNA in the blood.

________________________________________

Participants will:

* Receive the GC chemotherapy (gemcitabine and cisplatin) after having been treated with EVP
* Visit the clinic regularly for checkups, lab tests, and scans
* Answer questions about their health, quality of life, and daily function
* Provide blood samples for research

This study may help researchers find better ways to treat advanced bladder and urinary tract cancer in the future-especially for older adults or those who have already tried other treatments.

DETAILED DESCRIPTION:
This is a non-randomized single arm, two stage, open-label phase 2 efficacy study in adult patients with locally advanced or metastatic urothelial cancer. Subjects must have had one prior line of therapy consisting of EVP and have RECIST measurable disease prior to study entry. Patients will be treated with standard of care doses of all the chemotherapeutic drugs. Each cycle will consist of gemcitabine 1,000 mg/m2 administered over 30 minutes IV on days 1 and 8, followed by carboplatin AUC 5 on day 1, every 3 weeks. Patients will be treated until disease progression or any of the conditions listed in the protocol applies. Response to treatment will be evaluated by investigator determined CT scan or MRI every 9 weeks and the tumor will be assessed using RECIST v1.1 criteria. The study will be analyzed for futility after treatment of 19 patients. Patients who are not evaluable for the primary endpoint will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic or locally advanced histologically and radiographically confirmed urothelial carcinoma
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v1.1
* Patients must have received treatment with enfortumab vedotin plus pembrolizumab in the first line setting. Study treatment may be started within 28 days of last treatment with EV-P or with continuing toxicities if considered by the Sponsor-Investigator to be safe and within the best interest of the patient.
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have normal organ and marrow function as defined below.

  * Absolute neutrophil count > 1,000/mm3 unless patient has constitutional neutropenia
  * Platelets > 80,000/ul
  * Hemoglobin > 8.0 g/dL
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN or <3.5 x upper limit of normal (ULN) if liver metastases
  * Creatinine Clearance >20 mL/min
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* Optional: Archival tumor biospecimen, when available, must be procured for correlative evaluation. If tumor tissue is not available or accessible despite good faith efforts, patient may still be treated on study. Formalin fixed paraffin embedded (FFPE) tissue block(s) or at least 15 unbaked, unstained slides are required. Tissue samples taken from a metastatic lesion prior to the start of screening are acceptable.

Exclusion Criteria:

* Patients who have had systemic treatment including EV-P or radiotherapy within 2 weeks prior to entering the study
* Patients who have had systemic treatment including EV-P or radiotherapy within 2 weeks prior to entering the study
* Patients who have received more than one line of prior therapy or prior platinum-based chemotherapy for locally advanced or metastatic urothelial carcinoma (neoadjuvant platinum-based therapy including cisplatin is allowed)
* Patients who have not recovered from adverse events to less than Grade 2 secondary to agents administered more than 2 weeks prior to treatment initiation.
* Patients may not be receiving any other investigational agents
* Patients with uncontrolled and untreated CNS metastases:

  * Prior radiation to central nervous system (CNS) metastases is permitted
  * Prior history of CNS disease that has responded to previous systemic therapy is permitted only if no recurrence
  * Patient should not have leptomeningeal disease
  * CNS metastases have been clinically stable for at least 6 weeks prior to screening and baseline scans show no evidence of new or enlarged metastases
* Uncontrolled intercurrent illness including, but not limited to ongoing or active untreated infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit adherence with study requirements
* Subjects with a history of another invasive malignancy within 3 years before the first dose of study drug that cannot be watched and requires tumor- directed treatment, or any evidence of residual disease from a previously diagnosed malignancy that cannot be watched and requires treatment (adjuvant hormonal therapy for breast cancer is allowed)
* Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of chemotherapy (routine antimicrobial prophylaxis is permitted)
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Best overall response (Complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) to gemcitabine plus carboplatin defined per RECIST v 1.1 | 3 years
  From the start of the treatment until disease progression/recurrence

SECONDARY OUTCOMES:
To evaluate progression free survival (PFS) as a function of time since study enrollment in patients receiving GC after prior exposure to EVP | 3 years
  From initiation of study treatment until progression or death with patients who are still alive and progression free at the end of the follow-up period considered censored at their last contact.
To evaluate overall survival (OS) as a function of time since study enrollment in patients receiving GC after prior exposure to EVP | 3 years
  From initiation of study treatment until death with patients still alive at the end of follow-up censored at their last contact date
To evaluate the frequency and severity of toxicities attributed to GC after prior exposure to EVP | 3 years
  From the start of study treatment until the patient either begins survival follow-up, starts a new cancer therapy, or die, whichever occurs first
To evaluate the disease control rate (DCR) of gemcitabine plus carboplatin after prior exposure to EVP | 3 years
  From initiation of study treatment until progression or death with patients who are still alive and progression free at the end of the follow-up period considered censored at their last contact

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Geynisman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital at Broad Street, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No